CLINICAL TRIAL: NCT02974218
Title: Saint Luc Valve Registry
Acronym: SaLVaRe
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: Salvare
Record Dates: First submitted 2016-11-18; First posted 2016-11-28 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Valvular Heart Disease Stenosis and Regurgitation (Diagnosis)
MeSH Terms: conditions — Gastroesophageal Reflux; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The "Cliniques Universitaires Saint Luc" are one of the high specialized center in valvular heart diseases and valvular heart surgery. Aortic stenosis, mitral and aortic regurgitation are the three valve pathology that are mainly frequent and studied.

International guidelines in the management of valvular heart diseases are based on few limited old studies, mainly retrospective. And, a matter of concern is staying, about the timing of surgery for asymptomatic patients.

A prospective registry will help us to better understand the pathologies and try to better define guidelines criteria for surgery.

DETAILED DESCRIPTION:
With this prospective registry, all patients with aortic stenosis, mitral and aortic regurgitation will be followed. The investigators will find followed patients not yet operated or until surgery, but also patient after surgery according to the presence or abscence of guidelines criteria.

It will permit to compare different kind of management of patients with valvular heart disease and to better define guidelines criteria for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Presence of aortic stenosis, mitral or aortic regurgitation at the time of an echocardiography at the "Cliniques Universitaires Saint Luc".

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with valvular heart disease who undergo an echocardiography at the Cliniques Universitaires Saint Luc.
  Patients included must be > 18y and < 100 of age.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2000-01; Primary Completion 2020-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | every two years up to 10 years
  From the date of the first echocardiography until the date of death from any cause, documented progression and surgery will be regularly assessed up to 10 years.

CONTACTS AND LOCATIONS:
Overall Officials: Vanoverschlde Jean-Louis, MD, PhD, Study Director — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint Luc - Université Catholique de Louvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Clavel MA, Tribouilloy C, Vanoverschelde JL, Pizarro R, Suri RM, Szymanski C, Lazam S, Oberti P, Michelena HI, Jaffe A, Enriquez-Sarano M. Association of B-Type Natriuretic Peptide With Survival in Patients With Degenerative Mitral Regurgitation. J Am Coll Cardiol. 2016 Sep 20;68(12):1297-307. doi: 10.1016/j.jacc.2016.06.047. PMID 27634121
- [Result] Rezzoug N, Vaes B, de Meester C, Degryse J, Van Pottelbergh G, Mathei C, Adriaensen W, Pasquet A, Vanoverschelde JL. The clinical impact of valvular heart disease in a population-based cohort of subjects aged 80 and older. BMC Cardiovasc Disord. 2016 Jan 12;16:7. doi: 10.1186/s12872-016-0184-8. PMID 26754575
- [Result] de Meester C, Gerber BL, Vancraeynest D, Pouleur AC, Noirhomme P, Pasquet A, El Khoury G, Vanoverschelde JL. Early surgical intervention versus watchful waiting and outcomes for asymptomatic severe aortic regurgitation. J Thorac Cardiovasc Surg. 2015 Nov;150(5):1100-8. doi: 10.1016/j.jtcvs.2015.07.053. Epub 2015 Jul 28. PMID 26298872
- [Result] Rezzoug N, Vaes B, Pasquet A, Gerber B, de Meester C, Van Pottelbergh G, Adriaensen W, Mathei C, DeGryse J, Vanoverschelde JL. Prevalence and Prognostic Impact of Valve Area-Gradient Patterns in Patients >/=80 Years With Moderate-to-Severe Aortic Stenosis (from the Prospective BELFRAIL Study). Am J Cardiol. 2015 Sep 15;116(6):925-32. doi: 10.1016/j.amjcard.2015.05.062. Epub 2015 Jun 26. PMID 26219495
- [Result] Tribouilloy C, Rusinaru D, Charles V, Boulif J, Maes F, Levy F, Pasquet A, Marechaux S, Vanoverschelde JL. Progression of Low-Gradient, Low-Flow, Severe Aortic Stenosis With Preserved Left Ventricular Ejection Fraction. Am J Cardiol. 2015 Aug 15;116(4):612-7. doi: 10.1016/j.amjcard.2015.05.023. Epub 2015 May 21. PMID 26089012
- [Result] de Kerchove L, Mastrobuoni S, Boodhwani M, Astarci P, Rubay J, Poncelet A, Vanoverschelde JL, Noirhomme P, El Khoury G. The role of annular dimension and annuloplasty in tricuspid aortic valve repair. Eur J Cardiothorac Surg. 2016 Feb;49(2):428-37; discussion 437-8. doi: 10.1093/ejcts/ezv050. Epub 2015 Feb 26. PMID 25721823
- [Result] Barone-Rochette G, Pierard S, De Meester de Ravenstein C, Seldrum S, Melchior J, Maes F, Pouleur AC, Vancraeynest D, Pasquet A, Vanoverschelde JL, Gerber BL. Prognostic significance of LGE by CMR in aortic stenosis patients undergoing valve replacement. J Am Coll Cardiol. 2014 Jul 15;64(2):144-54. doi: 10.1016/j.jacc.2014.02.612. PMID 25011718
- [Result] Maes F, Boulif J, Pierard S, de Meester C, Melchior J, Gerber B, Vancraeynest D, Pouleur AC, Lazam S, Pasquet A, Vanoverschelde JL. Natural history of paradoxical low-gradient severe aortic stenosis. Circ Cardiovasc Imaging. 2014 Jul;7(4):714-22. doi: 10.1161/CIRCIMAGING.113.001695. Epub 2014 Apr 28. PMID 24777938
- [Result] de Meester C, Pasquet A, Gerber BL, Vancraeynest D, Noirhomme P, El Khoury G, Vanoverschelde JL. Valve repair improves the outcome of surgery for chronic severe aortic regurgitation: a propensity score analysis. J Thorac Cardiovasc Surg. 2014 Nov;148(5):1913-20. doi: 10.1016/j.jtcvs.2014.02.010. Epub 2014 Feb 10. PMID 24656668
- [Result] Pierard S, de Meester C, Seldrum S, Pasquet A, Gerber B, Vancraeynest D, Robert A, El Khoury G, Noirhomme P, Vanoverschelde JL. Impact of preoperative symptoms on postoperative survival in severe aortic stenosis: implications for the timing of surgery. Ann Thorac Surg. 2014 Mar;97(3):803-9. doi: 10.1016/j.athoracsur.2013.08.059. Epub 2013 Nov 5. PMID 24200400
- [Result] Barone-Rochette G, Pierard S, Seldrum S, de Meester de Ravenstein C, Melchior J, Maes F, Pouleur AC, Vancraeynest D, Pasquet A, Vanoverschelde JL, Gerber BL. Aortic valve area, stroke volume, left ventricular hypertrophy, remodeling, and fibrosis in aortic stenosis assessed by cardiac magnetic resonance imaging: comparison between high and low gradient and normal and low flow aortic stenosis. Circ Cardiovasc Imaging. 2013 Nov;6(6):1009-17. doi: 10.1161/CIRCIMAGING.113.000515. Epub 2013 Oct 7. PMID 24100045
- [Result] de Kerchove L, Boodhwani M, Glineur D, Vandyck M, Vanoverschelde JL, Noirhomme P, El Khoury G. Valve sparing-root replacement with the reimplantation technique to increase the durability of bicuspid aortic valve repair. J Thorac Cardiovasc Surg. 2011 Dec;142(6):1430-8. doi: 10.1016/j.jtcvs.2011.08.021. Epub 2011 Sep 28. PMID 21955470
- [Result] Pierard S, Seldrum S, de Meester C, Pasquet A, Gerber B, Vancraeynest D, El Khoury G, Noirhomme P, Robert A, Vanoverschelde JL. Incidence, determinants, and prognostic impact of operative refusal or denial in octogenarians with severe aortic stenosis. Ann Thorac Surg. 2011 Apr;91(4):1107-12. doi: 10.1016/j.athoracsur.2010.12.052. Epub 2011 Feb 18. PMID 21310391
- [Result] Boodhwani M, de Kerchove L, Watremez C, Glineur D, Vanoverschelde JL, Noirhomme P, El Khoury G. Assessment and repair of aortic valve cusp prolapse: implications for valve-sparing procedures. J Thorac Cardiovasc Surg. 2011 Apr;141(4):917-25. doi: 10.1016/j.jtcvs.2010.12.006. Epub 2011 Feb 3. PMID 21292284
- [Result] le Polain de Waroux JB, Pouleur AC, Robert A, Pasquet A, Gerber BL, Noirhomme P, El Khoury G, Vanoverschelde JL. Mechanisms of recurrent aortic regurgitation after aortic valve repair: predictive value of intraoperative transesophageal echocardiography. JACC Cardiovasc Imaging. 2009 Aug;2(8):931-9. doi: 10.1016/j.jcmg.2009.04.013. PMID 19679280
- [Result] Montant P, Chenot F, Robert A, Vancraeynest D, Pasquet A, Gerber B, Noirhomme P, El Khoury G, Vanoverschelde JL. Long-term survival in asymptomatic patients with severe degenerative mitral regurgitation: a propensity score-based comparison between an early surgical strategy and a conservative treatment approach. J Thorac Cardiovasc Surg. 2009 Dec;138(6):1339-48. doi: 10.1016/j.jtcvs.2009.03.046. Epub 2009 Jun 26. PMID 19660385
- [Result] Chenot F, Montant P, Vancraeynest D, Pasquet A, Gerber B, Noirhomme PH, El Khoury G, Vanoverschelde JL. Long-term clinical outcome of mitral valve repair in asymptomatic severe mitral regurgitation. Eur J Cardiothorac Surg. 2009 Sep;36(3):539-45. doi: 10.1016/j.ejcts.2009.02.063. Epub 2009 Jul 25. PMID 19632855
- [Result] Pouleur AC, le Polain de Waroux JB, Goffinet C, Vancraeynest D, Pasquet A, Gerber BL, Vanoverschelde JL. Accuracy of the flow convergence method for quantification of aortic regurgitation in patients with central versus eccentric jets. Am J Cardiol. 2008 Aug 15;102(4):475-80. doi: 10.1016/j.amjcard.2008.04.011. Epub 2008 May 24. PMID 18678309